CLINICAL TRIAL: NCT00344305
Title: A Phase 2, Open-Label, Single Arm Trial to Evaluate the Shedding and Safety of CAIV-T Administered to Children 6 to Less Than 60 Months of Age
Brief Title: A Study to Evaluate the Shedding and Safety of Trivalent Influenza Virus Vaccine Live, Intranasal in Infants and Young Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MI-CP129
Record Dates: First submitted 2006-06-22; First posted 2006-06-26 (Estimated); Results first posted 2010-11-01 (Estimated); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Healthy
Keywords: children, FluMist, shedding,
MeSH Terms: conditions — Influenza, Human | interventions — FluMist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Participants Between 6 to < 24 Months Age (Experimental): Participants received a single, intranasal dose of 0.2 millilitre (mL) (approximately 0.1 mL in each nostril) FluMist trivalent influenza virus vaccine live on Day 0 of the study. Each dose of FluMist vaccine contained 10^7 fluorescent focus units (FFU) of three influenza virus strains namely, A/New Caledonia/20/99 (H1N1), A/Wyoming/03/2003 (H3N2) (A/Fujian/411/2002-like) and B/Jilin/20/2003 (B/Shanghai/361/2002-like).
  Interventions: Biological: Trivalent influenza virus vaccine live, intranasal
- Cohort 2: Participants Between 24 to < 60 Months Age (Experimental): Participants received a single, intranasal dose of 0.2 mL (approximately 0.1 mL in each nostril) FluMist trivalent influenza virus vaccine live on Day 0 of the study. Each dose of FluMist vaccine contained 10^7 FFU of three influenza virus strains namely, A/New Caledonia/20/99 (H1N1), A/Wyoming/03/2003 (H3N2) (A/Fujian/411/2002-like) and B/Jilin/20/2003 (B/Shanghai/361/2002-like).
  Interventions: Biological: Trivalent influenza virus vaccine live, intranasal

INTERVENTIONS:
Biological: Trivalent influenza virus vaccine live, intranasal — A single, intranasal dose of 0.2 mL (approximately 0.1 mL in each nostril) FluMist trivalent influenza virus vaccine live on Day 0 of the study. Each dose of FluMist vaccine contained 10^7 FFU of three influenza virus strains.
  Other Names: FluMist; Cold-adapted influenza virus vaccine, trivalent (CAIV-T); Live attenuated influenza virus (LAIV)

SUMMARY:
Open label, single arm, multicenter study of the shedding and safety of a single dose of trivalent, influenza virus vaccine live, intranasal in children 6 to < 60 months of age, with 28-day shedding follow-up and 180-day safety follow-up.

DETAILED DESCRIPTION:
This was a Phase 2, open-label, single-arm, multicenter study designed to evaluate vaccine virus shedding and safety of trivalent influenza virus vaccine live, intranasal in children 6 to < 60 months of age. Enrollment of approximately 200 participants was stratified by age, with 100 participants 6 to < 24 months of age (who reached their sixth month but not their second year birthday) and 100 participants 24 to < 60 months of age (who reached their second year but not their fifth year birthday). Baseline medical history data collection included the participants prior receipt of influenza vaccine or history of laboratory-confirmed influenza illness in the previous influenza season.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 6 months to less than 60 months of age (reached their 6th month but not yet reached their 5th year birthday) at the time of study vaccination
* Written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization obtained from the participants parent/legal representative
* Ability of the participants parent/legal representative to understand and comply with the requirements of the study
* Participants parent/legal representative available by telephone
* Ability to complete follow-up period of 180 days after study vaccination as required by the protocol

Exclusion Criteria:

* History of hypersensitivity to any component of trivalent influenza virus vaccine live, intranasal, including egg or egg products, monosodium glutamate, or porcine gelatin
* History of hypersensitivity to gentamicin
* History of Guillain-Barré syndrome
* Medically diagnosed wheezing, bronchodilator use, or steroid use (systemic or inhaled), by parent/legal representative report or chart review, within the 42 days prior to study vaccination (i.e., children with recent persistent asthma were excluded); or history of severe persistent asthma according to the criteria described in the National Asthma Education and Prevention Program (NAEPP) Expert Panel Report
* Acute febrile (greater than or equal to [>=] 100.0 degree Fahrenheit [°F] oral or equivalent) and/or clinically significant respiratory illness (e.g., cough or sore throat) within 72 hours prior to study vaccination
* Any known immunosuppressive condition or immune deficiency disease (including human immunodeficiency virus [HIV] infection), or ongoing receipt of any immunosuppressive therapy
* Household contact who was immunocompromised (participants were also to avoid close contact with immunocompromised individuals for at least 21 days after study vaccination)
* Use of aspirin or aspirin-containing products within the 30 days prior to study vaccination, or expected receipt through 180 days after study vaccination
* Use of anti-influenza medications (including amantadine, rimantadine, oseltamivir, and zanamivir) within the 14 days prior to study vaccination, or expected receipt through 28 days after study vaccination
* Use of any intranasal medication within the 14 days prior to study vaccination, or expected receipt through 28 days after study vaccination
* Administration of any live virus vaccine within the 30 days prior to study vaccination, or expected receipt through 30 days after study vaccination
* Administration of any inactivated (i.e., non-live) vaccine within the 14 days prior to study vaccination, or expected receipt through 14 days after study vaccination
* Receipt of any investigational agent within the 30 days prior to study vaccination, or expected receipt through 180 days after study vaccination (use of licensed agents for indications not listed in the package insert was permitted)
* Receipt of any blood product within the 90 days prior to study vaccination, or expected receipt through 28 days after study vaccination
* Family member or household contact who was an employee of the research center or otherwise involved with the conduct of the study
* Any condition that in the opinion of the investigator would have interfered with evaluation of the vaccine or interpretation of study results

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2006-05-01 (Actual); Primary Completion 2006-07-01 (Actual); Study Completion 2006-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raburn Mallory, M.D., Study Director — MedImmune LLC
Locations (16):
- United States (16):
  - Little Rock Allergy & Asthma Clinic, PA, Little Rock, Arkansas
  - Pediatric and Adolescent Medicine, PA (PAMPA), Marietta, Georgia
  - Kentucky Pediatrics/Adult Research, Bardstown, Kentucky
  - Benchmark Research, Metairie, Louisiana
  - Health Sciences Research Center, Cortland, New York
  - Health Sciences Research Center, Elmira, New York
  - Regional Clinical Research Inc., Endwell, New York
  - Grand Prairie Pediatrics & Allergy Clinic, Oklahoma City, Oklahoma
  - Primary Physicians Research , Inc, Pittsburgh, Pennsylvania
  - Med-Pro Research Inc., Houston, Texas
  - Central Texas Health Research, New Braunfels, Texas
  - Benchmark Research, San Angelo, Texas
  - Wee Care Pediatrics, Layton, Utah
  - Utah Valley Pediatrics, Provo, Utah
  - PI-Coor Clinical Research, LLC, Burke, Virginia
  - Advanced Pediatrics, Vienna, Virginia

REFERENCES:
- [Result] Mallory RM, Yi T, Ambrose CS. Shedding of Ann Arbor strain live attenuated influenza vaccine virus in children 6-59 months of age. Vaccine. 2011 Jun 10;29(26):4322-7. doi: 10.1016/j.vaccine.2011.04.022. Epub 2011 Apr 20. PMID 21513761

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 200 participants were enrolled in the study from 15-May-2006 through 22-Jun-2006 at 16 sites in the United States of America.
Pre-assignment Details: A total of 200 participants were stratified on the basis of their age into two cohorts: Cohort 1 (participants aged between 6 to less than [<] 24 months) and Cohort 2 (participants aged between 24 to < 60 months).
Groups:
- Cohort 1: Participants Between 6 to < 24 Months Age: Participants received a single, intranasal dose of 0.2 millilitre (mL) (approximately 0.1 mL in each nostril FluMist trivalent influenza virus vaccine live on Day 0 of the study. Each dose of FluMist vaccine contained 10^7 fluorescent focus units (FFU) of three influenza virus strains namely, A/New Caledonia/20/99 (H1N1), A/Wyoming/03/2003 (H3N2) (A/Fujian/411/2002-like) and B/Jilin/20/2003 (B/Shanghai/361/2002-like).
Period: Overall Study
Arm/Group | Cohort 1: Participants Between 6 to < 24 Months Age | Cohort 2: Participants Between 24 to < 60 Months Age
Started | 100 | 100
Completed | 98 | 99
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Participant was not contacted in window | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Participants Between 6 to < 24 Months Age | Cohort 2: Participants Between 24 to < 60 Months Age | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: months] | 14.87 (5.50) | 41.31 (9.98) | 28.09 (15.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 53 | 104
  Male | 49 | 47 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 15 | 22
  Not Hispanic or Latino | 93 | 85 | 178
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 7 | 21
  White | 86 | 89 | 175
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
History of laboratory-confirmed influenza illness in previous influenza season [Number; unit: participants]
  Yes | 1 | 2 | 3
  No | 99 | 98 | 197
History of receiving an influenza vaccine [Number; unit: participants]
  Yes | 43 | 73 | 116
  No | 57 | 27 | 84

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Shed Any Vaccine Virus
Description: Viral shedding is defined as the detection of virus by viral culture and vaccine-type virus was confirmed by polymerase chain reaction (PCR) based assays. Viral shedding (A/New Caledonia/20/99 [H1N1]; A/Wyoming/03/2003 [H3N2] (A/Fujian/411/2002-like); B/Jilin/20/2003 B/Shanghai/361/2002-like]) was measured from samples obtained from nasal swabs daily from Days 1 to 7 post vaccination and approximately every other day thereafter from Days 9 to 28. Participants whose Day 25 or 28 shedding sample was positive for vaccine virus had additional shedding samples collected approximately every 7 days, or as soon as possible upon awareness of culture positivity, until 2 consecutive samples were negative for vaccine virus.
Time Frame: Days 1-28 after study vaccination (up to Day 28)
Population: Shedding population included all participants who received a full dose of study drug and had assay results from nasal specimens obtained at any post-dosing time point. Here, number of participants analyzed signified those participants who were evaluable for this outcome.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Participants Between 6 to < 24 Months Age | Cohort 2: Participants Between 24 to < 60 Months Age
Number analyzed (Participants) | 99 | 100
percentage of participants | 88.9 [81.0 to 94.3] | 69.0 [59.0 to 77.9]

2. Primary Outcome: Percentage of Participants Who Shed A/H1N1 Vaccine Virus
Description: Viral shedding is defined as the detection of virus by viral culture and vaccine-type virus was confirmed by PCR based assays. Viral shedding (A/New Caledonia/20/99 [H1N1]; A/Wyoming/03/2003 [H3N2] (A/Fujian/411/2002-like); B/Jilin/20/2003 B/Shanghai/361/2002-like]) was measured from samples obtained from nasal swabs daily from Days 1 to 7 post vaccination and approximately every other day thereafter from Days 9 to 28. Participants whose Day 25 or 28 shedding sample was positive for vaccine virus had additional shedding samples collected approximately every 7 days, or as soon as possible upon awareness of culture positivity, until 2 consecutive samples were negative for vaccine virus.
Time Frame: Days 1-28 after study vaccination (up to Day 28)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Participants Between 6 to < 24 Months Age | Cohort 2: Participants Between 24 to < 60 Months Age
Number analyzed (Participants) | 99 | 100
percentage of participants | 76.8 [67.2 to 84.7] | 52.0 [41.8 to 62.1]

3. Primary Outcome: Percentage of Participants Who Shed A/H3N2 Vaccine Virus
Description: as for outcome 2
Time Frame: Days 1-28 after study vaccination (up to Day 28)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Participants Between 6 to < 24 Months Age | Cohort 2: Participants Between 24 to < 60 Months Age
Number analyzed (Participants) | 99 | 100
percentage of participants | 57.6 [47.2 to 67.5] | 15.0 [8.6 to 23.5]

4. Primary Outcome: Percentage of Participants Who Shed B Vaccine Virus
Description: as for outcome 2
Time Frame: Days 1-28 after study vaccination (up to Day 28)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Participants Between 6 to < 24 Months Age | Cohort 2: Participants Between 24 to < 60 Months Age
Number analyzed (Participants) | 99 | 100
percentage of participants | 37.4 [27.9 to 47.7] | 37.0 [27.6 to 47.2]

5. Secondary Outcome: Duration of Any Vaccine Virus Shedding
Description: The number of days of shedding was summarized for all participants who shed any vaccine virus.
Time Frame: Days 1-28 after study vaccination (up to Day 28)
Population: Shedding population included all participants who received a full dose of study drug and had assay results from nasal specimens obtained at any post-dosing time point. Here, number of participants analyzed signified those participants who shed any confirmed strain virus.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Cohort 1: Participants Between 6 to < 24 Months Age | Cohort 2: Participants Between 24 to < 60 Months Age
Number analyzed (Participants) | 88 | 69
days | 3.0 (1.5) | 2.7 (1.6)

6. Secondary Outcome: Duration of Confirmed A/H1N1 Vaccine Virus Shedding
Description: The number of days of shedding was summarized for all participants who shed confirmed A/H1N1 strain virus.
Time Frame: Days 1-28 after study vaccination (up to Day 28)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Cohort 1: Participants Between 6 to < 24 Months Age | Cohort 2: Participants Between 24 to < 60 Months Age
Number analyzed (Participants) | 76 | 52
days | 2.1 (1.0) | 2.2 (1.3)

7. Secondary Outcome: Duration of Confirmed A/H3N2 Vaccine Virus Shedding
Description: The number of days of shedding was summarized for all participants who shed confirmed A/H3N2 strain virus.
Time Frame: Days 1-28 after study vaccination (up to Day 28)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Cohort 1: Participants Between 6 to < 24 Months Age | Cohort 2: Participants Between 24 to < 60 Months Age
Number analyzed (Participants) | 57 | 15
days | 1.8 (0.9) | 1.7 (0.8)

8. Secondary Outcome: Duration of Confirmed B Vaccine Virus Shedding
Description: The number of days of shedding was summarized for all participants who shed confirmed B strain virus.
Time Frame: Days 1-28 after study vaccination (up to Day 28)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Cohort 1: Participants Between 6 to < 24 Months Age | Cohort 2: Participants Between 24 to < 60 Months Age
Number analyzed (Participants) | 37 | 37
days | 2.1 (1.5) | 1.8 (1.2)

9. Secondary Outcome: Quantitation of Confirmed A/H1N1 Shed Vaccine Virus on Any Day
Description: Quantitation of confirmed A/H1N1 shed vaccine virus was evaluated using the log transformed median tissue culture infectious dose (TCID50) per (/) millilitre (mL) for A/H1N1 vaccine strain and summarized for all participants who shed vaccine virus.
Time Frame: Days 1-28 after study vaccination (up to Day 28)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: log (TCID50)/mL
Arm/Group | Cohort 1: Participants Between 6 to < 24 Months Age | Cohort 2: Participants Between 24 to < 60 Months Age
Number analyzed (Participants) | 52 | 45
log (TCID50)/mL | 2.14 (0.98) | 2.62 (0.97)

10. Secondary Outcome: Quantitation of Confirmed A/H3N2 Shed Vaccine Virus on Any Day
Description: Quantitation of confirmed A/H3N2 shed vaccine virus was evaluated using the log (TCID50)/mL for A/H3N2 vaccine strain and summarized for all participants who shed vaccine virus.
Time Frame: Days 1-28 after study vaccination (up to Day 28)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: log (TCID50)/mL
Arm/Group | Cohort 1: Participants Between 6 to < 24 Months Age | Cohort 2: Participants Between 24 to < 60 Months Age
Number analyzed (Participants) | 24 | 5
log (TCID50)/mL | 1.59 (0.95) | 1.10 (0.53)

11. Secondary Outcome: Quantitation of Confirmed B Shed Vaccine Virus on Any Day
Description: Quantitation of confirmed B shed vaccine virus was evaluated using the log (TCID50)/mL for B vaccine strain and summarized for all participants who shed vaccine virus.
Time Frame: Days 1-28 after study vaccination (up to Day 28)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: log (TCID50)/mL
Arm/Group | Cohort 1: Participants Between 6 to < 24 Months Age | Cohort 2: Participants Between 24 to < 60 Months Age
Number analyzed (Participants) | 28 | 29
log (TCID50)/mL | 1.70 (1.09) | 1.24 (0.68)

12. Secondary Outcome: Number of Participants With Genotypic and Phenotypic Stability of A/H1N1 Shed Vaccine Virus
Description: The genetic and phenotypic stability of shed vaccine virus was evaluated by determination of genomic sequence and assessment of the cold-adapted (ca) and temperature-sensitive (ts) phenotypes. Viruses were considered ts if their titer at 39 degrees Celsius (°C) was at least two logs (100-fold) lower than their titer at 33°C. Viruses were considered ca if they replicated at 25°C to a titer that was no more than two logs (100-fold) lower than the titer at 33°C. After additional phenotypic and genotypic analyses, all evaluable samples retained the ca and ts phenotypes.
Time Frame: Days 1-28 after study vaccination (up to Day 28)
Population: Shedding population: all participants who received a full dose of study drug and had assay results from nasal specimens obtained at any post-dosing time point. Here, number of participants analyzed signified those participants who were evaluable for this outcome and "n" signified those participants who were evaluable for a specified category.
Measure: Number; unit: participants
Groups:
- All Participants: Participants between 6 to < 60 months age received a single, intranasal dose of 0.2 mL (approximately 0.1 mL in each nostril) FluMist trivalent influenza virus vaccine live on Day 0 of the study. Each dose of FluMist vaccine contained 10^7 FFU of three influenza virus strains namely, A/New Caledonia/20/99 (H1N1), A/Wyoming/03/2003 (H3N2) (A/Fujian/411/2002-like) and B/Jilin/20/2003 (B/Shanghai/361/2002-like).
Arm/Group | All Participants
Number analyzed (Participants) | 93
participants
  Genotypic Stability (n=0) | NA — Data not available because no participant was evaluable for the specified category.
  Phenotypic Stability (n=93) | 90

13. Secondary Outcome: Number of Participants With Genotypic and Phenotypic Stability of A/H3N2 Shed Vaccine Virus
Description: The genetic and phenotypic stability of shed vaccine virus was evaluated by determination of genomic sequence and assessment of the ca and ts phenotypes. Viruses were considered ts if their titer at 39°C was at least two logs (100-fold) lower than their titer at 33°C. Viruses were considered ca if they replicated at 25°C to a titer that was no more than two logs (100-fold) lower than the titer at 33°C. After additional phenotypic and genotypic analyses, all evaluable samples retained the ca and ts phenotypes.
Time Frame: Days 1-28 after study vaccination (up to Day 28)
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 39
participants
  Genotypic Stability (n=0) | NA — Data not available because no participant was evaluable for the specified category.
  Phenotypic Stability (n=39) | 37

14. Secondary Outcome: Number of Participants With Genotypic and Phenotypic Stability of B Shed Vaccine Virus
Description: The genetic and phenotypic stability of shed vaccine virus was evaluated by determination of genomic sequence and assessment of the ca and ts phenotypes. Viruses were considered ts if their titer at 37°C was at least two logs (100-fold) lower than their titer at 33°C. Viruses were considered ca if they replicated at 25°C to a titer that was no more than two logs (100-fold) lower than the titer at 33°C. After additional phenotypic and genotypic analyses, all evaluable samples retained the ca and ts phenotypes.
Time Frame: Days 1-28 after study vaccination (up to Day 28)
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 61
participants
  Genotypic Stability (n=33) | 33
  Phenotypic Stability (n=61) | 29

15. Secondary Outcome: Number of Participants With Reactogenicity Events (REs) and Adverse Events (AEs) Through 28 Days Post Vaccination
Description: REs were predefined solicited events that could potentially occur after vaccination. The REs for this study were fever, runny/stuffy nose, sore throat, cough, vomiting, headache, abdominal pain (stomach ache), muscle ache, chills, decreased activity level (lethargy), decreased appetite, and irritability. An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Time Frame: Days 0-28 after vaccination (up to Day 28)
Population: Safety population included all participants who received any study drug and had experienced any follow-up for safety.
Measure: Number; unit: participants
Arm/Group | Cohort 1: Participants Between 6 to < 24 Months Age | Cohort 2: Participants Between 24 to < 60 Months Age
Number analyzed (Participants) | 100 | 100
participants
  Any REs | 84 | 77
  AEs | 48 | 31

16. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Significant New Medical Conditions (SNMC) Through 180 Days Post Vaccination
Description: An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. An SNMC is defined as a newly diagnosed medical condition that was of a chronic, ongoing nature and was assessed by the investigator as medically significant. SNMCs included, but were not limited to, diabetes, asthma, autoimmune disease (lupus, rheumatoid arthritis), and neurological disease (epilepsy, autism).
Time Frame: Days 0-180 after vaccination (up to 6.5 months)
Population: Safety population included all participants who received any study drug and had experienced any follow-up for safety.
Measure: Number; unit: participants
Arm/Group | Cohort 1: Participants Between 6 to < 24 Months Age | Cohort 2: Participants Between 24 to < 60 Months Age
Number analyzed (Participants) | 100 | 100
participants
  SAEs | 1 | 0
  SNMC | 1 | 1

17. Secondary Outcome: Number of Participants With REs in Relation to Any Vaccine Virus Shedding
Description: REs were predefined solicited events that could potentially occur after vaccination. The REs for this study were fever, runny/stuffy nose, sore throat, cough, vomiting, headache, abdominal pain (stomach ache), muscle ache, chills, decreased activity level (lethargy), decreased appetite, and irritability.
Time Frame: Days 0-28 after study vaccination (up to Day 28)
Population: Safety population included all participants who received any study drug and had experienced any follow-up for safety. Here, number of participants analyzed signified those participants who had REs.
Measure: Number; unit: participants
Arm/Group | Cohort 1: Participants Between 6 to < 24 Months Age | Cohort 2: Participants Between 24 to < 60 Months Age
Number analyzed (Participants) | 83 | 77
participants | 75 | 55

ADVERSE EVENTS:
Time Frame: AEs - Days 0-28 post dosing (up to Day 28); SAEs - Days 0-180 post dosing (up to 6.5 months)
Arm/Group | Cohort 1: Participants Between 6 to < 24 Months Age | Cohort 2: Participants Between 24 to < 60 Months Age
Serious Adverse Events (participants affected / at risk) | 1/100 | 0/100
Other Adverse Events (participants affected / at risk) | 48/100 | 25/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Participants Between 6 to < 24 Months Age (N=100) | Cohort 2: Participants Between 24 to < 60 Months Age (N=100)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Participants Between 6 to < 24 Months Age (N=100) | Cohort 2: Participants Between 24 to < 60 Months Age (N=100)
OTORRHOEA (Ear and labyrinth disorders) | 2 (2) | 0 (0)
CONJUNCTIVITIS (Eye disorders) | 2 (2) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 5 (6) | 9 (11)
FLATULENCE (Gastrointestinal disorders) | 2 (4) | 0 (0)
TEETHING (Gastrointestinal disorders) | 21 (30) | 0 (0)
HERPANGINA (Infections and infestations) | 2 (2) | 0 (0)
OTITIS MEDIA (Infections and infestations) | 4 (4) | 0 (0)
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 1 (1) | 3 (3)
VIRAL INFECTION (Infections and infestations) | 3 (4) | 2 (2)
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
ARTHROPOD STING (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
BODY TEMPERATURE INCREASED (Investigations) | 3 (4) | 2 (2)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
ECZEMA (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
HEAT RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restricion is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.